CLINICAL TRIAL: NCT00201747
Title: Phase II Randomized Trial of Sequentially Administered CPT-11 and Mitomycin C in Patients With Advanced Esophageal and Stomach Cancer
Brief Title: Sequentially Administered CPT-11 and Mitomycin C in Patients With Advanced Esophageal and Stomach Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: Pharmacia and Upjohn (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-0151
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2017-12-06 (Actual); Status verified 2017-12

CONDITIONS: Esophageal Cancer; Esophagus Cancer; Cancer of Stomach; Stomach Cancer
Keywords: Advanced
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms | interventions — Irinotecan; Mitomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: CPT-11 — CPT-11 will be administered intravenously on days 2 and 9 (24 hours after MMC, when the MMC is required) Two weeks of rest (beginning days 15 and 22) (drug free) will complete the cycle, with therapy planned to be resumed on day 29.
Drug: Mitomycin C — MMC will be administered intravenously on day 1 (Arm A) and days 1 and 8 (Arm B)

SUMMARY:
To determine the most efficacious of two combination regimens of sequential CPT-11 and MMC in patients with advanced and previously untreated esophageal and GE junction adenocarcinomas.

DETAILED DESCRIPTION:
Rationale: Previous studies suggest that both irinotecan and Mytomycin C when administered alone have some efficacy against stomach cancer. Based on laboratory testing, researchers hypothesized that Mytomycin C may enhance the efficacy of irinotecan through an enzyme called Topoisomerase I. In addition, because Mytomycin C has severe side effects, combining these chemotherapy agents together may allow for lower dosages resulting in greater efficacy and reduced side effects. A recent study indicates that the combination of these drugs has promising anti-tumor activity against esophageal and stomach cancers. The current study builds on previous research to explore the most effective schedule for administering these drugs together.

Purpose: This study is evaluating the combination of irinotecan and Mytomycin C on two different treatment schedules in patients with advanced esophageal and stomach cancers. Characteristics of different genes will also be measured, along with genetic and molecular changes by comparing test results from the beginning and end of the study.

Treatment: Patients in this study will receive irinotecan and Mytomycin C in one of two treatment schedules. Both drugs will be administered in patients through an intravenous infusion. A computer will randomly assign patients to a treatment group. Group one will receive Mytomycin C on day 1 and irinotecan on days 2 and 9. Group two will receive Mytomycin C on days 1 and 8 and irinotecan on days 2 and 9. After day 9, patients in both groups will not be given any study drugs for almost three weeks to complete a four week cycle. Several tests and exams will be given throughout the study to closely monitor patients. Patients will continue receiving the study drugs until they experience disease growth or unacceptable side effects.

ELIGIBILITY:
Inclusion Criteria:

* Must have pathologically confirmed & measurable advanced esophageal or Gastroesophageal junction adenocarcinoma
* No prior chemotherapy
* Prior radiation allowed if <=20% of bone marrow was irradiated
* Target lesions must not be in radiation field.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2001-09; Primary Completion 2006-10 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Most efficacious of two combination regimens of sequential CPT-11 and MMC in patients with advanced and previously untreated esophageal and GE junction adenocarcinomas | 2001-2010

SECONDARY OUTCOMES:
Evaluate gene expression profile of NQ01, and Topo I genes in peripheral blood mononuclear cells and tumor tissue during therapy with MMC and CPT-11 | 2001-2010
Evaluate the frequency of NQ01 gene mutations in patients with esophageal and GE junction adenocarcinomas and its association to prognosis and antitumor activity. | 2001-2010
Evaluate if pre- and/or post-treatment Topo I-, CE and NQ01-gene expression in fresh tumor specimens and adjacent tissue, are associated with antitumor efficacy or toxicity. | 2001-2010

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Villalona, MD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University, Columbus, Ohio, United States

REFERENCES:
- [Result] Lustberg MB, Bekaii-Saab T, Young D, Otterson G, Burak W, Abbas A, McCracken-Bussa B, Lustberg ME, Villalona-Calero MA. Phase II randomized study of two regimens of sequentially administered mitomycin C and irinotecan in patients with unresectable esophageal and gastroesophageal adenocarcinoma. J Thorac Oncol. 2010 May;5(5):713-8. doi: 10.1097/JTO.0b013e3181d7776d. PMID 20354452
- See also: Jamesline — http://cancer.osu.edu